CLINICAL TRIAL: NCT05835063
Title: We Chatt (Communication, Hopes, Action, Tips and Team) A Study to Improve Physician-Youth Communication and Medical Decision Making
Brief Title: A Study to Improve Physician-Youth Communication and Medical Decision Making
Acronym: CHATT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Melissa Cousino, Associate Professor of Pediatrics, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00231699; 5K23HL145096-04 (NIH)
Record Dates: First submitted 2023-04-17; First posted 2023-04-28 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure NYHA Class II; Heart Failure NYHA Class III; Heart Failure NYHA Class IV
Keywords: Caregiver/parent
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: A total of 20 physicians will be recruited. 10 will be randomized to participate in the intervention arm and 10 will be randomized to the control arm. Participants and caretakers will account for approximately 60 enrolled participants that will not be randomized.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- We Chatt communication tool (Experimental)
  Interventions: Behavioral: We Chatt communication tool
- Usual care (Placebo Comparator)
  Interventions: Behavioral: Usual/standard care

INTERVENTIONS:
Behavioral: We Chatt communication tool — This arm involves the collaborative completion of a 2-page communication preferences document between a primary physician and an adolescent/young adult patient. Physicians will participate in a 1-hour training led by study principal investigator featuring didactic, multimedia, and experiential-based learning to support the facilitation of the WE CHATT intervention with patients.
  Arms: We Chatt communication tool
Behavioral: Usual/standard care — Usual/standard care will be provided. Physicians randomized to the control arm will not receive training in the WE CHATT communication intervention.
  Arms: Usual care

SUMMARY:
The goal of this study is improving patient-centered communication for young people with advanced heart disease.

ELIGIBILITY:
Physician Inclusion Criteria:

* Physician participants will be recruited from the Division of Pediatric Cardiology at the University of Michigan. All physicians with dedicated clinical effort will be eligible.
* Eligible physicians must anticipate remaining on staff >1 year

Patient/Caregiver Inclusion Criteria:

* Patients 12-24 years old with heart failure symptoms meeting criteria for New York Heart Association (NYHA) Class II - IV heart failure
* One parent/caregiver of patient participants meeting inclusion criteria will also be eligible

Physician Exclusion Criteria:

- Not a physician at University of Michigan in the Division of Pediatric Cardiology

Patient/Caregiver Exclusion Criteria:

* Patients with significant cognitive/developmental delay with potential to impact study participation will be excluded from the study due to the focus on physician-youth communication.
* Parents and parent/caregivers that are non-English speaking will be excluded from this pilot study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Cousino, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Clinician Intervention Arm: Clinicians who were randomized to this arm used the WE CHATT tool in communicating with patient participants. Clinician participants in this arm completed a 1-hour training to support their facilitation of the WE CHATT intervention with patients.
- Clinician Control Arm: Clinician participants in this arm did not receive training in the WE CHATT communication intervention. Usual/standard care was provided.
- Patients: Patient participants (12-24 years of age) with heart failure symptoms meeting criteria for New York Heart Association (NYHA) Class II - IV heart failure (i.e., limitations in physical activity, fatigue, palpitations, dyspnea).
- Parent Caregiver: One parent/caregiver of patient participants.
Period: Overall Study
Arm/Group | Clinician Intervention Arm | Clinician Control Arm | Patients | Parent Caregiver
Started | 10 | 10 | 10 | 9
Completed | 10 | 10 | 10 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinician Intervention Arm | Clinician Control Arm | Patients | Parent Caregiver | Total
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 39
Age, Categorical [Count of Participants; unit: Participants] — Population: Age data was not collected for participants in the Parent arm.
  Participants
    number analyzed (Participants) | 10 | 10 | 10 | 0 | 30
    <=18 years | 0 | 0 | 9 |  | 9
    Between 18 and 65 years | 10 | 10 | 1 |  | 21
    >=65 years | 0 | 0 | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 7 | 19
  Male | 6 | 6 | 6 | 2 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity data was not collected for participants in the Parent arm.
  Participants
    number analyzed (Participants) | 10 | 10 | 10 | 0 | 30
    Hispanic or Latino | 0 | 1 | 0 |  | 1
    Not Hispanic or Latino | 10 | 9 | 10 |  | 29
    Unknown or Not Reported | 0 | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 0 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 2
  White | 5 | 10 | 8 | 8 | 31
  More than one race | 1 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 10 | 9 | 39

OUTCOME MEASURES:

1. Primary Outcome: Physician Overall Satisfaction With the We Chatt Intervention Based on the Post Clinician Survey
Description: Satisfaction was based on the answers for 12 questions in which clinicians selected from a Likert scale from strongly disagree (1) -Strongly agree (5). The scores ranged from 12-60; higher scores indicated greater satisfaction.
Time Frame: 2 weeks (after intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Clinicians Intervention: Clinicians who were randomized to this arm used the WE CHATT tool in communicating with patient participants. Clinician participants in this arm completed a 1-hour training to support their facilitation of the WE CHATT intervention with patients.
Arm/Group | Clinicians Intervention
Number analyzed (Participants) | 10
score on a scale | 57.4 (2.7)

2. Primary Outcome: Patient/Caregiver Overall Satisfaction With the We Chatt Intervention Based on the Patient/Caregiver Survey
Description: Parent/Caregiver completed 12 questions in which participants selected from a Likert scale from Strongly disagree (1) to Strongly agree (5). The scores ranged from 12-60; higher scores indicated greater satisfaction.
Time Frame: 2 weeks (after intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Caregivers: One parent/caregiver of patient participants.
Arm/Group | Patients | Caregivers
Number analyzed (Participants) | 10 | 10
score on a scale | 49.5 (5.8) | 53.4 (5.2)

3. Secondary Outcome: Physician Satisfaction With the We Chatt Intervention From Physicians Based on the Post Clinician Survey
Description: Physicians answered 1 question on a scale from 0 to 10 (with 0 being worst and 10 being best)
Time Frame: 2 weeks (after intervention)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Clinicians Intervention
Number analyzed (Participants) | 10
score on a scale | 9 [9 to 9]

4. Secondary Outcome: Patient/Caregiver Satisfaction With the We Chatt Intervention Based on the Patient/Caregiver Survey
Description: Patient/Caregiver answered 1 question on a scale from 0 to 10 (with 0 being worst and 10 being best)
Time Frame: 2 weeks (after intervention)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Patients | Caregivers
Number analyzed (Participants) | 10 | 9
score on a scale | 9 [8 to 9] | 10 [9 to 10]

5. Secondary Outcome: Time (Measured in Minutes) to Complete We Chatt the Intervention by Clinicians
Description: Number of minutes to complete the intervention was collected on clinician survey.
Time Frame: 30 minutes (approximately)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Clinicians Intervention
Number analyzed (Participants) | 10
minutes | 15 [15 to 25]

ADVERSE EVENTS:
Time Frame: Up to 28 days
Arm/Group | Clinician Intervention Arm | Clinician Control Arm | Patients | Parent Caregiver
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT05835063/Prot_SAP_001.pdf
  • Informed Consent Form (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/63/NCT05835063/ICF_000.pdf